CLINICAL TRIAL: NCT01616758
Title: Phase II, Open Label Study to Examine Androgen Receptor Status and the Activity of GTx-024 Hormonal Therapy in Women With Estrogen Receptor Positive Metastatic Breast Cancer Who Have Previously Responded to Hormone Therapy
Brief Title: Phase II Study of GTx024 in Women With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G200801
Record Dates: First submitted 2012-06-07; First posted 2012-06-12 (Estimated); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ostarine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GTx-024 9mg (Experimental): GTx-024 dosage of three soft gels once daily to equal 9mg
  Interventions: Drug: GTx-024 9mg

INTERVENTIONS:
Drug: GTx-024 9mg
  Other Names: GTx-024 dosage of three soft gels once daily to equal 9mg

SUMMARY:
The primary efficacy analysis will be the clinical benefit at 6 months as measured by a modified Response Evaluation Criteria in Solid Tumors RECIST classification. Key secondary endpoints of objective response rate, progression free survival, time to progression, duration of response, effects on physical function, and effects on tumor progression in women with Androgen Receptor positive breast cancer will also be assessed.

DETAILED DESCRIPTION:
This is an open label, multicenter study to assess the safety and efficacy of GTx-024 in female subjects who have estrogen receptor (ER) positive metastatic breast cancer and who have responded previously to hormone therapy. Subjects may have received up to 3 prior hormonal therapies for the treatment of breast cancer. Subjects must have responded to adjuvant hormonal therapy for > 3 years or hormonal therapy for metastatic disease for > 6 months before progression to be eligible for this study.

The primary efficacy analysis will be the clinical benefit in subjects with AR positive breast cancer at 6 months as measured by a modified Response Evaluation Criteria In Solid Tumors (RECIST 1.1) classification. Key secondary endpoints of clinical benefit in all subjects and AR negative subjects, as well as objective response rate, progression free survival, time to progression, duration of response, incidence of SREs, and time to first SRE in subsets based on AR status will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Give voluntary, signed informed consent in accordance with institutional policies.
2. Be a woman that has been diagnosed with ER positive metastatic breast cancer.
3. Have metastatic breast cancer with measurable lesions prior to enrollment or bone only disease prior to enrollment. A measurable lesion is defined as one lesion whose longest diameter (LD) can be accurately measured as 10 mm CT or MRI technique by using a 5 mm contiguous reconstruction algorithm. Measurable lesions must be at least 2 times the slice thickness or at least two times the size of the CT scan interval cut. Patients with bone only disease and non-measurable lesions are eligible.
4. Be clinically confirmed as postmenopausal. Subjects must have undergone the onset of spontaneous, medical or surgical menopause prior to the start of this study.(Spontaneous menopause is defined as the natural cessation of ovarian function as indicated by being amenorrheic for at least 12 months. If the subject has been amenorrheic for > or equal to 6 months but < 12 months, they must have a serum FSH concentration of > or equal to 50 mIU/mL and an estradiol concentration of less than or equal to 25 pg/mL. Medical menopause is defined as treatment with a luteinizing hormone receptor hormone agonist and surgical menopause is defined as bilateral oophorectomy).
5. Have been treated and responded to previous adjuvant hormonal therapy for 3 years or previous hormonal therapy for metastatic disease for 6 months prior to disease progression.
6. Have not had radiation therapy for breast cancer within 2 weeks of randomization in this study and are not planned to have radiation therapy during participation in this study.
7. Be willing to provide a formalin-fixed, paraffin-embedded block(s) of cancerous tissue from a biopsy of a metastatic tumor lesion(s) collected during the two (2) years prior to study entry or as a component of enrollment in the study for determination of AR and ER status. Tissue samples from a biopsy of a primary tumor lesion will also be provided if available.
8. Serum creatinine 2.0 mg/dL
9. Have ECOG score 2.
10. Be age 18 years.

Exclusion Criteria:

1. Have triple negative breast cancer
2. Have, in the judgment of the Investigator, a clinically significant concurrent illness or psychological, familial, sociological, geographical or other concomitant condition that would not permit adequate follow-up and compliance with the study protocol
3. Have uncontrolled hypertension (systolic blood pressure greater than 150 mm Hg and/or diastolic blood pressure greater than 100 mm Hg despite treatment with antihypertensive drugs)
4. Untreated congestive heart failure or untreated angina
5. Have Stage 4 chronic obstructive pulmonary disease (COPD)
6. Have positive screen for Hepatitis B consisting of HBsAg (Hepatitis B Surface Antigen), unless subject was diagnosed > 10 years prior to enrollment and no evidence of active liver disease
7. The presence of consistently abnormal clinical laboratory test (Appendix B) values which are considered clinically significant. In addition, any subject with total bilirubin above 2 times the upper limit of normal (ULN) or liver enzymes ( ALT/SGOT or AST/SGPT) above 1.5 times the ULN without evidence of liver metastases or above 5 times the ULN in subjects with evidence of liver metastases will not be admitted to the study
8. Have positive screen for hepatitis A antibody IgM or HIV
9. Have received chemotherapy for metastatic breast cancer within the 3 months prior to enrollment in the study or be expected to receive chemotherapy for metastatic breast cancer during the study
10. Be currently taking testosterone, methyltestosterone, oxandrolone (Oxandrin®),oxymetholone, danazol, fluoxymesterone (Halotestin®), testosterone-like agents (such as dehydroepiandrosterone (DHEA), androstenedione, and other androgenic compounds, including herbals), or antiandrogens. Previous therapy with testosterone and testosterone-like agents is acceptable with a 30-day washout (if previous testosterone therapy was long term depot within the past 6 months, the site should contact the medical monitor (1-877-693-2723) for this study to determine appropriate washout period).
11. Have untreated or uncontrolled brain metastasis
12. Have been diagnosed with or treated for cancer within the previous two years, other than breast cancer or non-melanoma carcinoma of the skin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mayzie Johnston, PharmD, Study Director — GTx
Locations (4):
- United States (4):
  - AMPM Research Clinic, Miami, Florida
  - Illinois Cancer Care, PC, Peoria, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Commonwealth Hematology-Oncology, Lawrence, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- GTx-024 9mg: GTx-024 dosage of three soft gels once daily to equal 9mg
  GTx-024 9mg
Period: Overall Study
Arm/Group | GTx-024 9mg
Started | 22
Evaluable | 20
Completed | 0
Not Completed | 22
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Disease progression | 18
Not completed — Study termination by Sponsor | 1

BASELINE CHARACTERISTICS:
Population: All Enrolled patients Note: 20 patients were deemed as evaluable
Arm/Group | GTx-024 9mg
Number analyzed (Participants) | 22
Age, Customized [Count of Participants; unit: Participants]
  ≥18 years | 22
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Treated With GTx024 With Clinical Benefit With AR Positive Breast Cancer
Description: N=17 of 22 subjects with AR Positive Breast Cancer - Clinical Benefit is defined as a complete response (CR), partial response (PR), or stable disease (SD).
Time Frame: 6 months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | GTx-024 9mg
Number analyzed (Participants) | 17
Participants | 6

2. Secondary Outcome: Percentage of Subjects Treated With GTx024 With Clinical Benefit (All Subjects)
Description: Clinical Benefit is defined as a complete response (CR), partial response (PR), or stable disease (SD).
Time Frame: 6 Months
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | GTx-024 9mg
Number analyzed (Participants) | 22
Participants | 7

3. Secondary Outcome: Percentage of Subjects Treated With GTx024 Achieving Objective Response by 1 Year of Treatment
Description: Objective Response is defined as achieving Complete or Partial Response on Tumor Assessments
  Note: Due to zero subject achieving response, all subsequent outcome measures related to response cannot be conducted.
Time Frame: 1 Year
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | GTx-024 9mg
Number analyzed (Participants) | 22
Participants | 0

ADVERSE EVENTS:
Arm/Group | GTx-024 9mg
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 2/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GTx-024 9mg (N=22)
Pathologic Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain of Chest (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GTx-024 9mg (N=22)
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 4
Hot Flush (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No